CLINICAL TRIAL: NCT03700671
Title: The Effects of Low-Volume High Intensity Interval Training and Circuit Training on Maximal Oxygen Uptake
Brief Title: High Intensity Interval Training Versus Circuit Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Hull (Other)
Responsible Party: Principal Investigator, Stefan Birkett, Lecturer in Exercise Science, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UCentralLancashire
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: High Intensity Interval Training
MeSH Terms: interventions — High-Intensity Interval Training; Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: Participants were randomised to either high or moderate intensity exercise
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): HIIT was set at > 85% HRmax. Active recovery was set at 25-50 watts. Sessions were performed using cycle ergometry.
  Interventions: Other: High intensity interval training
- Circuit training (Active Comparator): The CT group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80%. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated. Each station was occupied for three to six minutes depending on session duration with minimal rest in-between.
  Interventions: Other: Circuit training

INTERVENTIONS:
Other: High intensity interval training — Participants performed HIIT twice a week for eight weeks. Findings were compared to moderate intensity continuous training which followed the same exercise frequency and duration
  Arms: High intensity interval training
Other: Circuit training — The CT group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80% HRmax twice per week for eight weeks. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated
  Arms: Circuit training

SUMMARY:
High intensity interval training (HIIT) and circuit training (CT) are popular methods of exercise, eliciting improvements in cardiorespiratory fitness (CRF). However direct comparisons of these two training methods are limited.

DETAILED DESCRIPTION:
Study Design Participants were enrolled in a randomised control trial at the University of Hull to either eight weeks of High intensity interval training (HIIT) or Circuit Training (CT) (two supervised sessions per week, accompanied by an exercise physiologist). A sample size of 38 using G Power 3.1 software was calculated based on previously published data in which the mean difference between HIIT and Moderate Intensity Continuous Training (MICT) was 3.2 ml.kg-1.min-1 with a pooled standard deviation of 3 ml.kg-1.min-1. Statistical significance was set at 0.05 and power set to 0.95. To allow for 10% attrition 42 individuals were recruited to the study. To assess the effectiveness of the interventions as determined by maximal oxygen consumption (VO2max), a maximal cardiopulmonary exercise test (CPET) to volitional exhaustion on an electronically braked cycle ergometer at baseline (visit one), and following an eight-week exercise intervention of HIIT or CT (visit two) was conducted. When attending the assessments participants were asked not to take part in any strenuous exercise 24 hours prior to the appointment, to wear suitable comfortable clothing and avoid a large meal. Visit two CPET was performed within six days of completing the exercise interventions. A thorough warm-up and cool down before and after each exercise session. All were asked to maintain their habitual physical activity patterns during the intervention. Body mass index (BMI) was calculated by dividing body weight by height in meters squared and was presented as kg.m-2. Resting blood pressure was measured after 15 minutes of rest using a sphygmomanometer (A.C. Cossor & Son Ltd, London UK) and stethoscope (3M Healthcare, St Paul, MN). To provide a comprehensive account of the study the Consensus on Exercise Reporting Template (CERT) was consulted.

Participants Ethical approval was provided by the School of Life Sciences ethics committee at the University of Hull which was in accordance with the 1964 Helsinki declaration and its later amendments or comparable ethical standards. A total of 42 apparently healthy men and women between the age of 18-65 years were recruited to the study. Enrolled individuals reported no medical history of cardiometabolic or limiting respiratory disease, were non-smokers, had a body mass index <30 kg.m-2, classified as recreationally active and none were taking any medication that would affect heart rate. As a condition of enrolment, those over 45 years obtained written medical clearance from a general practitioner and underwent resting and exercise 12-lead electrocardiogram (ECG) (GE Healthcare, Chalfont St Giles, United Kingdom). Written informed consent and a pre-exercise medical questionnaire was completed by all.

Cardiopulmonary Exercise Testing Maximal CPETs were conducted in accordance with the American Thoracic Society (ATS) and the American College of Chest Physicians (ACCP) guidelines. An Oxycon pro (Jaeger, Hoechburg, Germany) breath by breath metabolic cart was used to collect respiratory gas exchange data. Automatic and manual calibration evaluated ambient temperature, humidity, barometric pressure and altitude. Calibration of the air flow volume was conducted using a 3 litre syringe and by automatic calibration. Two-point gas calibration was also conducted to ensure accurate measures of inspired oxygen and expired carbon dioxide. Tests were performed on a GE e-bike ergometer (GE Healthcare, Buckinghamshire, UK) using a ramp protocol. The protocol consisted of a three-minute rest phase, three minutes of unloaded cycling, followed by a personalised ramp test (ramp rate ranged between 15 and 30 watts) with work rate continually increased every one to three seconds. Participants performed the same ramp rate pre and post testing. Participants were asked to pedal at a cadence of 70 rpm until they reached volitional exhaustion at a protocol duration between eight to twelve minutes. Self-reported rating of perceived exertion (RPE) scores using the 6-20 scale and heart rate (HR) (FT1 heart rate monitor, Polar Electro, Finland) was recorded during the last five seconds of each minute of the test, at maximum exercise and during the recovery period. Together with verbal encouragement to volitional exhaustion, VO2max was attained by participants achieving at least two of the following criteria, VO2 plateau as determined by a failure of VO2 increase by 150 ml/min with further increases in workload analysed by breath by breath gas exchange data averaged over 15 seconds, respiratory exchange ratio (RER) > 1.10, achieve > 85% age predicated heart rate maximum (HRmax) and a RPE > 17 on the 6-20 Borg scale. VO2 at the ventilatory anaerobic threshold (VAT) was defined using the V slope method and verified using ventilatory equivalents. Peak power output (PPO) (watts) and HRmax were defined as the highest value achieved during the CPET with maximum oxygen and heart rate (VO2 /HR) determined by the ratio of VO2max and HRmax.

Training Interventions The HIIT group were asked to perform ten one-minute HIIT intervals, each followed by one minute of active recovery (AR) (total exercise time 20 minutes). Resulting from the CPET, HIIT was set at above 85% HRmax with a specific HR designated for this criterion. Active recovery was set at a load corresponding to 25-50 watts. Sessions were performed on a Wattbike trainer (Wattbike Ltd, Nottingham, UK). The CT group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand/squats, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80% HRmax (calculated from CPET). No resistance equipment was involved, only body weight. Participants initially performed 20 minutes of CT with duration increased by five minutes per week until the desired 40 minutes. Each station was occupied for three to six minutes depending on session duration, moving from one station to the next with minimal rest. During both interventions, HR was measured in last 5 seconds of each station/interval using a FT1 polar heart rate monitor (Polar Electro, Finland) with each CT session timed using a stop watch (Axprod S.L, Guipuzcoa, Spain). Intensity for both interventions was adjusted throughout by the investigator to ensure an appropriate HR range and successful completion of the protocol. Participants were made aware of their HR ranges and verbal encouragement was given by the physiologist to help achieve and maintain these thresholds. Energy expenditure between HIIT and CT was not matched.

To assess the validity of the exercise interventions, participant fidelity to the desired exercise intensity was determined using cut points of >85% HRmax and 60-80% HRmax for HIIT and CT respectively and reported using previous examples. These values were calculated using the participants mean heart rate for each individual interval or station over the 16 sessions and was expressed as a percentage of HRmax as determined by CPET at visit 1. Specific fidelity thresholds were consulted to determine low (<50%), moderate (50-70%) and high (>70%) compliance. Adherence was determined as a percentage of completed sessions, with 14 (> 85%) being the threshold for completion.

Statistical Analysis Statistical analysis was conducted using Statistical Package for the Social Sciences (SPSS) version 24 (IBM, New York, USA). An independent t-test was used to identify group differences at baseline. Assumptions of normality were verified using the Shapiro-Wilk test. Skewness and kurtosis of distribution was visually examined. Non-normally distributed data was presented as median and interquartile range (IQR). A two-way (condition x time) repeated measures analysis of variance (ANOVA) was used to compare CRF pre-and post-training. Post-hoc analysis for the main effects and interactions was assessed using a Bonferroni adjustment. Group differences were compared using independent t tests. Variables were displayed as mean with 95% confidence intervals (95% CI) or standard deviation where specified. Partial eta squared effect sizes were also calculated with 0.01, 0.06 and 0.14 representing small, medium and large effect sizes, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Participants reported no medical history of cardiometabolic or limiting respiratory disease, were non-smokers, had a body mass index <30 kg.m-2, classified as recreationally active

Exclusion Criteria:

* Cardiometabolic disease, high activity levels, Unable to tolerate the exercise intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Birkett, PhD, Principal Investigator — University of Central Lancashire
Locations (1):
- Univeristy of Hull, Hull, Kingston Upon Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross R, Blair SN, Arena R, Church TS, Despres JP, Franklin BA, Haskell WL, Kaminsky LA, Levine BD, Lavie CJ, Myers J, Niebauer J, Sallis R, Sawada SS, Sui X, Wisloff U; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Cardiovascular and Stroke Nursing; Council on Functional Genomics and Translational Biology; Stroke Council. Importance of Assessing Cardiorespiratory Fitness in Clinical Practice: A Case for Fitness as a Clinical Vital Sign: A Scientific Statement From the American Heart Association. Circulation. 2016 Dec 13;134(24):e653-e699. doi: 10.1161/CIR.0000000000000461. Epub 2016 Nov 21. PMID 27881567
- [Background] Kaminsky LA, Arena R, Beckie TM, Brubaker PH, Church TS, Forman DE, Franklin BA, Gulati M, Lavie CJ, Myers J, Patel MJ, Pina IL, Weintraub WS, Williams MA; American Heart Association Advocacy Coordinating Committee, Council on Clinical Cardiology, and Council on Nutrition, Physical Activity and Metabolism. The importance of cardiorespiratory fitness in the United States: the need for a national registry: a policy statement from the American Heart Association. Circulation. 2013 Feb 5;127(5):652-62. doi: 10.1161/CIR.0b013e31827ee100. Epub 2013 Jan 7. No abstract available. PMID 23295916
- [Background] Lee DC, Artero EG, Sui X, Blair SN. Mortality trends in the general population: the importance of cardiorespiratory fitness. J Psychopharmacol. 2010 Nov;24(4 Suppl):27-35. doi: 10.1177/1359786810382057. PMID 20923918
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Background] Weston M, Taylor KL, Batterham AM, Hopkins WG. Effects of low-volume high-intensity interval training (HIT) on fitness in adults: a meta-analysis of controlled and non-controlled trials. Sports Med. 2014 Jul;44(7):1005-17. doi: 10.1007/s40279-014-0180-z. PMID 24743927
- [Background] Taylor KL, Weston M, Batterham AM. Evaluating intervention fidelity: an example from a high-intensity interval training study. PLoS One. 2015 Apr 22;10(4):e0125166. doi: 10.1371/journal.pone.0125166. eCollection 2015. PMID 25902066
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] McGregor G, Nichols S, Hamborg T, Bryning L, Tudor-Edwards R, Markland D, Mercer J, Birkett S, Ennis S, Powell R, Begg B, Haykowsky MJ, Banerjee P, Ingle L, Shave R, Backx K. High-intensity interval training versus moderate-intensity steady-state training in UK cardiac rehabilitation programmes (HIIT or MISS UK): study protocol for a multicentre randomised controlled trial and economic evaluation. BMJ Open. 2016 Nov 16;6(11):e012843. doi: 10.1136/bmjopen-2016-012843. PMID 27852718
- [Background] Esfandiari S, Sasson Z, Goodman JM. Short-term high-intensity interval and continuous moderate-intensity training improve maximal aerobic power and diastolic filling during exercise. Eur J Appl Physiol. 2014 Feb;114(2):331-43. doi: 10.1007/s00421-013-2773-x. Epub 2013 Nov 27. PMID 24281825
- [Background] Sawyer BJ, Tucker WJ, Bhammar DM, Ryder JR, Sweazea KL, Gaesser GA. Effects of high-intensity interval training and moderate-intensity continuous training on endothelial function and cardiometabolic risk markers in obese adults. J Appl Physiol (1985). 2016 Jul 1;121(1):279-88. doi: 10.1152/japplphysiol.00024.2016. Epub 2016 Jun 2. PMID 27255523
- [Background] Baekkerud FH, Solberg F, Leinan IM, Wisloff U, Karlsen T, Rognmo O. Comparison of Three Popular Exercise Modalities on V O2max in Overweight and Obese. Med Sci Sports Exerc. 2016 Mar;48(3):491-8. doi: 10.1249/MSS.0000000000000777. PMID 26440134
- [Background] Boyd JC, Simpson CA, Jung ME, Gurd BJ. Reducing the intensity and volume of interval training diminishes cardiovascular adaptation but not mitochondrial biogenesis in overweight/obese men. PLoS One. 2013 Jul 5;8(7):e68091. doi: 10.1371/journal.pone.0068091. Print 2013. PMID 23861854
- [Background] Stavrinou PS, Bogdanis GC, Giannaki CD, Terzis G, Hadjicharalambous M. High-intensity Interval Training Frequency: Cardiometabolic Effects and Quality of Life. Int J Sports Med. 2018 Feb;39(3):210-217. doi: 10.1055/s-0043-125074. Epub 2018 Feb 2. PMID 29396978
- [Background] Hood MS, Little JP, Tarnopolsky MA, Myslik F, Gibala MJ. Low-volume interval training improves muscle oxidative capacity in sedentary adults. Med Sci Sports Exerc. 2011 Oct;43(10):1849-56. doi: 10.1249/MSS.0b013e3182199834. PMID 21448086
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Slade SC, Dionne CE, Underwood M, Buchbinder R. Consensus on Exercise Reporting Template (CERT): Explanation and Elaboration Statement. Br J Sports Med. 2016 Dec;50(23):1428-1437. doi: 10.1136/bjsports-2016-096651. Epub 2016 Oct 5. PMID 27707738
- [Background] Ross RM. ATS/ACCP statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 May 15;167(10):1451; author reply 1451. doi: 10.1164/ajrccm.167.10.950. No abstract available. PMID 12738602
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Nordestgaard BG, Chapman MJ, Ray K, Boren J, Andreotti F, Watts GF, Ginsberg H, Amarenco P, Catapano A, Descamps OS, Fisher E, Kovanen PT, Kuivenhoven JA, Lesnik P, Masana L, Reiner Z, Taskinen MR, Tokgozoglu L, Tybjaerg-Hansen A; European Atherosclerosis Society Consensus Panel. Lipoprotein(a) as a cardiovascular risk factor: current status. Eur Heart J. 2010 Dec;31(23):2844-53. doi: 10.1093/eurheartj/ehq386. Epub 2010 Oct 21. PMID 20965889
- [Background] Richardson JTE. Eta squared and partial eta squared as measures of effect size in educational research. Educational Research Review. 2011;6(2):135-47. doi:https://doi.org/10.1016/j.edurev.2010.12.001.
- [Background] Matsuo T, Saotome K, Seino S, Eto M, Shimojo N, Matsushita A, Iemitsu M, Ohshima H, Tanaka K, Mukai C. Low-volume, high-intensity, aerobic interval exercise for sedentary adults: VO(2)max, cardiac mass, and heart rate recovery. Eur J Appl Physiol. 2014 Sep;114(9):1963-72. doi: 10.1007/s00421-014-2917-7. Epub 2014 Jun 11. PMID 24917354
- [Background] Ingle L, Mellis M, Brodie D, Sandercock GR. Associations between cardiorespiratory fitness and the metabolic syndrome in British men. Heart. 2017 Apr;103(7):524-528. doi: 10.1136/heartjnl-2016-310142. Epub 2016 Oct 25. PMID 27798054
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] Currie KD, Dubberley JB, McKelvie RS, MacDonald MJ. Low-volume, high-intensity interval training in patients with CAD. Med Sci Sports Exerc. 2013 Aug;45(8):1436-42. doi: 10.1249/MSS.0b013e31828bbbd4. PMID 23470301
- [Background] McKay BR, Paterson DH, Kowalchuk JM. Effect of short-term high-intensity interval training vs. continuous training on O2 uptake kinetics, muscle deoxygenation, and exercise performance. J Appl Physiol (1985). 2009 Jul;107(1):128-38. doi: 10.1152/japplphysiol.90828.2008. Epub 2009 May 14. PMID 19443744
- [Background] Montero D, Lundby C. Refuting the myth of non-response to exercise training: 'non-responders' do respond to higher dose of training. J Physiol. 2017 Jun 1;595(11):3377-3387. doi: 10.1113/JP273480. Epub 2017 May 14. PMID 28133739
- [Background] Bhambhani Y, Norris S, Bell G. Prediction of stroke volume from oxygen pulse measurements in untrained and trained men. Can J Appl Physiol. 1994 Mar;19(1):49-59. doi: 10.1139/h94-003. PMID 8186762
- [Background] Daussin FN, Ponsot E, Dufour SP, Lonsdorfer-Wolf E, Doutreleau S, Geny B, Piquard F, Richard R. Improvement of VO2max by cardiac output and oxygen extraction adaptation during intermittent versus continuous endurance training. Eur J Appl Physiol. 2007 Oct;101(3):377-83. doi: 10.1007/s00421-007-0499-3. Epub 2007 Jul 28. PMID 17661072
- [Background] Little JP, Safdar A, Wilkin GP, Tarnopolsky MA, Gibala MJ. A practical model of low-volume high-intensity interval training induces mitochondrial biogenesis in human skeletal muscle: potential mechanisms. J Physiol. 2010 Mar 15;588(Pt 6):1011-22. doi: 10.1113/jphysiol.2009.181743. Epub 2010 Jan 25. PMID 20100740
- [Background] Astorino TA, Edmunds RM, Clark A, King L, Gallant RA, Namm S, Fischer A, Wood KM. High-Intensity Interval Training Increases Cardiac Output and V O2max. Med Sci Sports Exerc. 2017 Feb;49(2):265-273. doi: 10.1249/MSS.0000000000001099. PMID 27669447
- [Background] Helgerud J, Hoydal K, Wang E, Karlsen T, Berg P, Bjerkaas M, Simonsen T, Helgesen C, Hjorth N, Bach R, Hoff J. Aerobic high-intensity intervals improve VO2max more than moderate training. Med Sci Sports Exerc. 2007 Apr;39(4):665-71. doi: 10.1249/mss.0b013e3180304570. PMID 17414804
- [Background] Ziemann E, Grzywacz T, Luszczyk M, Laskowski R, Olek RA, Gibson AL. Aerobic and anaerobic changes with high-intensity interval training in active college-aged men. J Strength Cond Res. 2011 Apr;25(4):1104-12. doi: 10.1519/JSC.0b013e3181d09ec9. PMID 20661160
- [Background] Astorino TA, deRevere J, Anderson T, Kellogg E, Holstrom P, Ring S, Ghaseb N. Change in VO2max and time trial performance in response to high-intensity interval training prescribed using ventilatory threshold. Eur J Appl Physiol. 2018 Sep;118(9):1811-1820. doi: 10.1007/s00421-018-3910-3. Epub 2018 Jun 19. PMID 29923111
- [Background] Ghosh AK. Anaerobic threshold: its concept and role in endurance sport. Malays J Med Sci. 2004 Jan;11(1):24-36. PMID 22977357
- [Background] Fortington LV, Donaldson A, Lathlean T, Young WB, Gabbe BJ, Lloyd D, Finch CF. When 'just doing it' is not enough: assessing the fidelity of player performance of an injury prevention exercise program. J Sci Med Sport. 2015 May;18(3):272-7. doi: 10.1016/j.jsams.2014.05.001. Epub 2014 May 16. PMID 24930985
- [Background] Tucker WJ, Sawyer BJ, Jarrett CL, Bhammar DM, Gaesser GA. Physiological Responses to High-Intensity Interval Exercise Differing in Interval Duration. J Strength Cond Res. 2015 Dec;29(12):3326-35. doi: 10.1519/JSC.0000000000001000. PMID 25970496
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- [Background] Ciolac EG, Mantuani SS, Neiva CM, Verardi C, Pessoa-Filho DM, Pimenta L. Rating of perceived exertion as a tool for prescribing and self regulating interval training: a pilot study. Biol Sport. 2015 Jun;32(2):103-8. doi: 10.5604/20831862.1134312. Epub 2015 Jan 15. PMID 26028809
- [Background] Blair SN, Morris JN. Healthy hearts--and the universal benefits of being physically active: physical activity and health. Ann Epidemiol. 2009 Apr;19(4):253-6. doi: 10.1016/j.annepidem.2009.01.019. PMID 19344864
- [Background] Blair SN, Kohl HW 3rd, Paffenbarger RS Jr, Clark DG, Cooper KH, Gibbons LW. Physical fitness and all-cause mortality. A prospective study of healthy men and women. JAMA. 1989 Nov 3;262(17):2395-401. doi: 10.1001/jama.262.17.2395. PMID 2795824
- [Background] Hardcastle SJ, Ray H, Beale L, Hagger MS. Why sprint interval training is inappropriate for a largely sedentary population. Front Psychol. 2014 Dec 23;5:1505. doi: 10.3389/fpsyg.2014.01505. eCollection 2014. No abstract available. PMID 25566166
- [Background] Weston M, Batterham AM, Tew GA, Kothmann E, Kerr K, Nawaz S, Yates D, Danjoux G. Patients Awaiting Surgical Repair for Large Abdominal Aortic Aneurysms Can Exercise at Moderate to Hard Intensities with a Low Risk of Adverse Events. Front Physiol. 2017 Jan 9;7:684. doi: 10.3389/fphys.2016.00684. eCollection 2016. PMID 28119627
- [Background] Hurst C, Weston KL, Weston M. The effect of 12 weeks of combined upper- and lower-body high-intensity interval training on muscular and cardiorespiratory fitness in older adults. Aging Clin Exp Res. 2019 May;31(5):661-671. doi: 10.1007/s40520-018-1015-9. Epub 2018 Jul 26. PMID 30051418

RESULTS

PARTICIPANT FLOW:
Groups:
- High Intensity Interval Training: High intensity interval training (HIIT) was set at > 85% HRmax. Active recovery was set at 25-50 watts. Sessions were performed using cycle ergometry.
  High intensity interval training: Participants performed HIIT twice a week for eight weeks. Findings were compared to moderate intensity continuous training which followed the same exercise frequency and duration
- Circuit Training: The Circuit Training (CT) group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80%. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated. Each station was occupied for three to six minutes depending on session duration with minimal rest in-between.
  Circuit training: The CT group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80% HRmax twice per week for eight weeks. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated
Period: Overall Study
Arm/Group | High Intensity Interval Training | Circuit Training
Started | 21 | 21
Completed | 20 | 19
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 2

BASELINE CHARACTERISTICS:
Population: no race or ethnicity exclusion
Groups:
- High Intensity Interval Training: Perform High intensity interval training twice per week for 8 weeks
- Circuit Training: Perform Circuit training twice per week for 8 weeks
- Total: Total of all reporting groups
Arm/Group | High Intensity Interval Training | Circuit Training | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (12.3) | 41.2 (12.9) | 41.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 21 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 19 | 39
Body mass index [Mean (Standard Deviation); unit: kg.m-2] | 24.4 (2.3) | 25.9 (2.7) | 25.2 (2.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 122 (14) | 126 (11) | 124 (12)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 75 (11) | 79 (9) | 77 (10)
Resting heart rate [Mean (Standard Deviation); unit: bpm] | 68 (12) | 67 (10) | 68 (11)
Respiratory exchange ratio at VO2max [Mean (Standard Deviation); unit: unitless] | 1.30 (0.12) | 1.31 (0.12) | 1.31 (0.12)
Heart rate maximum [Mean (Standard Deviation); unit: bpm] | 174 (12) | 174 (14) | 174 (13)
Maximum oxygen consumption/heart rate [Mean (Standard Deviation); unit: ml.beat-1] | 12.8 (3.7) | 13.9 (3.9) | 13.6 (3.8)
Peak power output [Mean (Standard Deviation); unit: watts] | 191.9 (43.7) | 209.8 (55.2) | 200.9 (49.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximal Oxygen Consumption (ml.Kg-1.Min-1)
Description: Maximal oxygen consumption (ml.kg-1.min-1), as determined during a cardiopulmonary exercise test (CPET) represents the upper limit of aerobic fitness in humans. A low VO2max is associated with a greater risk of premature all-cause and cardiovascular mortality, independent of traditional risk factors and physical activity status. Conversely, increasing VO2max through exercise training may improve cardiometabolic health, quality of life and increase life-expectancy
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Groups:
- High Intensity Interval Training: High intensity interval training was set at > 85% HRmax. Active recovery was set at 25-50 watts. Sessions were performed using cycle ergometry.
  High intensity interval training: Participants performed HIIT twice a week for eight weeks. Findings were compared to moderate intensity continuous training which followed the same exercise frequency and duration
- Circuit Training: The circuit training group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80%. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated. Each station was occupied for three to six minutes depending on session duration with minimal rest in-between.
  Circuit training: The CT group completed a practical seven-station mixed modality exercise circuit (cycle ergometer, rower, treadmill, sit to stand, knee to elbow and leg kickback with bicep curl) at an intensity of 60-80% HRmax twice per week for eight weeks. Participants initially performed 20 minutes of CT with duration gradually increased to the desired 40 minutes as tolerated
Arm/Group | High Intensity Interval Training | Circuit Training
Number analyzed (Participants) | 20 | 19
ml/kg/min
  Pre Intervention | 31.5 (7.1) | 31.4 (6.8)
  Post Intervention | 35.4 (7.3) | 32.4 (6.2)
Statistical Analysis 1: Comparison: High Intensity Interval Training vs Circuit Training; A sample size of 38 using G*Power 3.1 software was calculated based on previously published data in which the mean difference between HIIT and moderate intensity continuous training (MICT) was 3.2 ml.kg-1.min-1 with a pooled standard deviation of 3 ml.kg-1.min-1. Statistical significance was set at = 0.05 and power set to 0.95. To allow for 10% attrition 42 individuals were recruited to the study; Test type: Superiority; p < 0.01, ANOVA — A P-value of 0.05 was used as the threshold for significance

2. Secondary Outcome: Oxygen Consumption at the Ventilatory Anaerobic Threshold
Description: Oxygen consumption at the Ventilatory Anaerobic Threshold ml/kg/min. This measure will assess if individuals can exercise at higher intensities before lactate accumulation, thus becoming 'physiologically efficient
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | High Intensity Interval Training | Circuit Training
Number analyzed (Participants) | 20 | 19
ml/kg/min
  Pre Intervention | 15.5 (2.7) | 15.6 (3.0)
  Post Intervention | 17.9 (2.5) | 16.2 (3.1)
Statistical Analysis 1: Comparison: High Intensity Interval Training vs Circuit Training; Test type: Superiority; p < 0.01, ANOVA — 0.05 was used as a threshold for significance

3. Other Pre Specified Outcome: Intervention Fidelity - Participants That Complied With the Exercise Protocols
Description: To assess if the interventions were delivered as intended, percentage of participants that complied with the exercise protocols
Time Frame: 8 weeks
Population: To assess the validity of the exercise interventions, participant fidelity to the desired exercise intensity was determined using cut points using specific cut points. Fidelity was measured over the course of the 16 sessions.
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | High Intensity Interval Training | Circuit Training
Number analyzed (Participants) | 20 | 19
Percentage | 90 [80 to 100] | 86 [76 to 96]

4. Other Pre Specified Outcome: The Percentage of Individuals That Responsed to the Intervention
Description: If participants had a postive increased in maximal oxygen consumption following the two interventions
Time Frame: 8 weeks
Population: A percentage of participants that increased maximal oxygen consumption
Measure: Number; unit: Percentage
Arm/Group | High Intensity Interval Training | Circuit Training
Number analyzed (Participants) | 20 | 19
Percentage | 100 | 78

ADVERSE EVENTS:
Time Frame: Data was collected for each participant over the course of their intervention which was 8 weeks
Arm/Group | High Intensity Interval Training | Circuit Training
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03700671/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03700671/Prot_SAP_001.pdf